CLINICAL TRIAL: NCT04274218
Title: Locomotor Response of Persons With Upper Limb Loss to Treadmill Perturbations
Brief Title: Upper Limb Loss Perturbation Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3290-P; 1I21RX003290-01A1 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Amputation
Keywords: Stability; Locomotion; Motor Control; Trip; Falls; Upper Limb Loss; Prosthesis; Arm

STUDY DESIGN:
Intervention Model Description: Participants will receive a small treadmill belt disturbance while walking.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walking perturbation - Free (Experimental): Healthy controls without limb loss and individuals with upper limb loss between the wrist and elbow will receive a treadmill belt disturbance while walking. Able-bodied individuals will walk with both arms free and individuals with amputation will walk with their prosthesis.
  Interventions: Other: Perturbation
- Walking perturbation - Limited (Experimental): Healthy controls without limb loss and individuals with upper limb loss between the wrist and elbow will receive a treadmill belt disturbance while walking. Able-bodied individuals will walk with one arm bound to their side with straps and individuals with amputation will walk without their prosthesis.
  Interventions: Other: Perturbation

INTERVENTIONS:
Other: Perturbation — Participants from both cohorts will experience a simulated trip while walking on the treadmill. The trip is induced through a rapid acceleration and deceleration of the treadmill belt speed.

SUMMARY:
Recent investigations have suggested that persons with upper limb loss experience a high prevalence of falls with a quarter of reported falls resulting from a trip. Moreover, studies indicate that missing part of an arm may negatively impact balance and that use of a prosthesis exacerbates this problem. While the investigators are beginning to understand the effects of upper limb loss on balance, the understanding of how Veterans with upper limb loss respond to walking disturbances is incomplete. Therefore, the aims of this study are to observe the effects of upper limb loss and wearing a prosthesis on the preparation and recovery of Veterans who trip during walking. The investigators plan to use unique treadmill technology to deliver controlled, yet unexpected, perturbations to Veterans with upper limb loss and non-amputee controls, and assess walking stability through body dynamics. Results from this study will help us understand why Veterans with upper limb loss fall as a critical first step to addressing this problem through balance-targeted interventions that are integrated into patient care.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to characterize the proactive and reactive locomotor response of Veterans with upper limb loss (ULL) to a trip during walking. The investigators' recent VA-funded investigations have suggested that persons with ULL experience a high prevalence of falls and demonstrate postural control mechanisms that may impair stability. Specifically, nearly half of individuals with ULL at or proximal to the wrist level experience at least one fall per year and almost a third will experience two or more falls. Further, use of a prosthesis increases the likelihood of falling by six times, 25% of reported falls resulted from tripping, and nearly a third of individuals who experience a fall suffer a fall-related injury. Falls can have considerable economic burden on the VHA and lead to long-term diminished quality of life. The investigators' biomechanical studies suggest that persons with unilateral ULL display greater postural sway during standing than able-bodied individuals which increases when wearing a prosthesis, and right/left asymmetry in locomotor stability dynamics that may increase the risk of falling toward the impaired limb side and during sound limb side strides. These findings emphasize the need for additional research to better understand the mechanisms Veterans with ULL use to control balance and how wearing a prosthesis affects these strategies. As the investigators' previous research was concerned with steady-state characterization of postural control, the investigators now plan to build on this work by studying the effects of ULL and wearing a prosthesis on locomotor stability when responding to a trip disturbance during walking. In this context, locomotor stability is defined as the ability to recover from a perturbation and return to steady-state gait.

The investigators will address the study aims by analyzing trip-induced proactive and reactive locomotor strategy differences in two study comparisons: 1) Veterans with unilateral transradial level ULL against matched able-bodied controls (with and without one arm bound), and 2) Veterans with unilateral transradial ULL when wearing their customary prosthesis against not wearing their prosthesis. Controlled, yet unexpected, simulated trips will be delivered through the investigators' custom-built treadmill which permits programmable belt velocity disturbances and allows participants to continue walking following recovery. The investigators will characterize the proactive and reactive locomotor stability mechanisms through a set of biomechanical (angular momentum, arm and trunk kinematics) variables. Biomechanical variables will be quantified using an optical motion capture system. The investigators expect that Veterans with ULL will demonstrate altered locomotor stability mechanisms compared to controls, and these differences will exist between wearing and not wearing their customary prosthesis. Results from this study will help us characterize the underlying mechanisms of locomotor stability in Veterans with ULL and identify the factors associated with their increased prevalence of trip-related falls. Such knowledge is a critical first step to addressing this public health problem through stability-targeted rehabilitation interventions aimed at reducing falls, fall-related injuries, and associated VHA costs in this Veteran patient group. The investigators will use the outcomes from this pilot study to guide future VA Merit Award proposals to develop and assess physical training intervention methods and wearable and prosthetic technology to improve stability in Veterans with ULL. The VHA is an ideal venue to pursue this work as one of its main priorities is to elevate the standard-of-care for Veterans with limb loss.

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion criteria for all participants include:

* age between 18 and 65 years
* normal or corrected vision
* able to walk unassisted for 20 minutes without undue fatigue or health risks

Additional inclusion criteria for participants with ULL include:

* unilateral ULL at the transradial level
* most recent major upper limb amputation occurred at least one year prior to study
* residuum and amputated side in good condition (no scars, infections, pain, etc.)
* habitual experience using an upper limb prosthesis for at least one year
* a self-reported comfortable prosthetic suspension

Exclusion Criteria:

Exclusion criteria for all participants include:

* self-reported additional neurological, vascular, or musculoskeletal pathologies (other than ULL when applicable) that may affect proprioception/balance
* self-reported medication that may affect proprioception/balance, e.g.:

  * drugs that are ototoxic, such as certain Aminoglycosides and pain killers
* cognitive deficits that preclude understanding of the study instructions
* presence of osteoporosis
* presence of pacemakers or stents that may be irritated by the chest harness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Major, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants with upper limb absence and 10 healthy controls were screened for eligibility between December 1 2020 and February 10 2022. Individuals with upper limb loss were recruited from clinics providing prosthetics care and education programs for prosthetics. Healthy controls were recruited from the Chicago community.
Pre-assignment Details: All 20 participants agreed to participate and completed the study protocol.
Groups:
- Healthy Controls - Arms Free Then One Arm Bound; Healthy Controls - One Arm Bound Then Both Arms Free: Healthy controls without limb loss provided demographic information, then completed baseline walking for 1 minute, and then received a treadmill belt disturbance while walking under two conditions in a cross-over study design. Healthy controls either walked with both arms free first, then with one arm bound, OR with one arm bound first, then with both arms free. The order of arms free and bound conditions were randomized. There is no washout period and each condition lasted for 15 minutes.
- Upper Limb Absence - With Prosthesis First Then w/o Prosthesis; Upper Limb Absenece - w/o Prosthesis First Then With Prosthesis: Individuals with upper limb loss between the wrist and elbow provided demographic information, then completed baseline walking for 1 minute, and then received a treadmill belt disturbance while walking while walking under two conditions in a cross-over study design. Individuals with upper limb loss walked either with their prosthesis first, then without their prosthesis, OR without their prosthesis first, then with their prosthesis. The order of with and without prosthesis conditions were randomized. There is no washout period and each condition lasted for 15 minutes.
Period: Demographic Information (10 Minutes)
Arm/Group | Healthy Controls - Arms Free Then One Arm Bound | Upper Limb Absence - With Prosthesis First Then w/o Prosthesis | Healthy Controls - One Arm Bound Then Both Arms Free | Upper Limb Absenece - w/o Prosthesis First Then With Prosthesis
Started | 5 | 6 | 5 | 4
Completed | 5 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Baseline Walking (1 Minute)
Arm/Group | Healthy Controls - Arms Free Then One Arm Bound | Upper Limb Absence - With Prosthesis First Then w/o Prosthesis | Healthy Controls - One Arm Bound Then Both Arms Free | Upper Limb Absenece - w/o Prosthesis First Then With Prosthesis
Started | 5 | 6 | 5 | 4
Completed | 5 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Perturbation Condition 1 (15 Minutes)
Arm/Group | Healthy Controls - Arms Free Then One Arm Bound | Upper Limb Absence - With Prosthesis First Then w/o Prosthesis | Healthy Controls - One Arm Bound Then Both Arms Free | Upper Limb Absenece - w/o Prosthesis First Then With Prosthesis
Started | 5 | 6 | 5 | 4
Completed | 5 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Perturbation Condition 1 (15 Minutes)
Arm/Group | Healthy Controls - Arms Free Then One Arm Bound | Upper Limb Absence - With Prosthesis First Then w/o Prosthesis | Healthy Controls - One Arm Bound Then Both Arms Free | Upper Limb Absenece - w/o Prosthesis First Then With Prosthesis
Started | 5 | 6 | 5 | 4
Completed | 5 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy controls and individuals with unilateral transradial limb absence
Groups:
- Healthy Controls: Healthy controls without limb loss will receive a treadmill belt disturbance while walking. Able-bodied individuals will walk with both arms free and with one arm bound.
- Upper Limb Absence: Individuals with upper limb loss between the wrist and elbow will receive a treadmill belt disturbance while walking with and without their prosthesis.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Upper Limb Absence | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (16) | 44 (15) | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 9 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Whole-body Angular Momentum in Sagittal-plane; Momentum of the Body in the Sagittal Plane of Walking Progression
Description: Whole-body angular momentum is the momentum of all limb segments about the Body Center of Mass (BCoM) summed. Whole-body angular momentum is estimated in the sagittal plane, which is the plane of walking progression, and the range of this value is normalized to a person's body mass, height, and walking speed. Whole body angular momentum is minimized by the central nervous system to facilitate postural control. For this study, whole body angular momentum range was averaged across the 12 perturbation trials and then across all participants. To note, the reported whole body angular momentum values are the relative increase from baseline to perturbation recovery that are all measured in the same session. There are no additional sessions as the baseline whole body angular momentum reflects those values before the perturbation trials.
Time Frame: 1 hour
Population: Data collected for each participant during baseline and when recovering from the perturbation.
Measure: Mean (Standard Deviation); unit: Unitless (normalized)
Groups:
- Healthy Controls Arms Free: Healthy controls with both arms free to move.
- Upper Limb Absence Without Prosthesis: Individuals with upper limb absence not wearing their prosthesis.
- Healthy Controls One Arm Bound: Healthy controls with the non-dominant arm bound to the body.
- Upper Limb Absence With Prosthesis: Individuals with upper limb absence wearing their prosthesis.
Arm/Group | Healthy Controls Arms Free | Upper Limb Absence Without Prosthesis | Healthy Controls One Arm Bound | Upper Limb Absence With Prosthesis
Number analyzed (Participants) | 10 | 10 | 10 | 10
Unitless (normalized) | 0.025 (0.0006) | 0.031 (0.006) | 0.027 (0.009) | 0.028 (0.006)

2. Secondary Outcome: Shoulder Angle Flexion-extension Range
Description: Range-of-motion for shoulder joint angle flexion-extension of the impaired or non-dominant arm (Deg) during perturbation recovery; Dynamics used for postural control to regulate and reduce whole-body angular momentum during trip response.
Time Frame: 1 hour
Population: Range of motion of shoulder flexion-extension of the impaired (individuals with upper limb absence) or non-dominant arm (healthy controls) during perturbation recovery.
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Healthy Controls With Arms Free: Healthy controls with both arms free to move.
- Healthy Controls With One Arm Bound: Healthy controls with the non-dominant arm bound to the body.
Arm/Group | Healthy Controls With Arms Free | Upper Limb Absence Without Prosthesis | Healthy Controls With One Arm Bound | Upper Limb Absence With Prosthesis
Number analyzed (Participants) | 10 | 10 | 10 | 10
Degrees | 36 (18) | 34 (10) | 5 (1) | 31 (16)

3. Secondary Outcome: Trunk Flexion Angle
Description: Maximum flexion angle (degrees) of the trunk during perturbation recovery.
Time Frame: 1 hour
Population: Controls with both arms free or one arm bound and persons with upper limb absence wearing or not wearing their prosthesis.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Healthy Controls With Arms Free | Upper Limb Absence Without Prosthesis | Healthy Controls With One Arm Bound | Upper Limb Absence With Prosthesis
Number analyzed (Participants) | 10 | 10 | 10 | 10
Degrees | 9.9 (3.1) | 10.1 (2.7) | 10.1 (4.1) | 10.2 (2.7)

4. Secondary Outcome: Trunk Flexion Velocity
Description: Maximum trunk flexion velocity (deg/s) during perturbation recovery
Time Frame: 1 hour
Population: Controls with both arms free or one arm bound and persons with upper limb absence with or without their prosthesis.
Measure: Mean (Standard Deviation); unit: Degrees/second
Arm/Group | Healthy Controls With Arms Free | Upper Limb Absence Without Prosthesis | Healthy Controls With One Arm Bound | Upper Limb Absence With Prosthesis
Number analyzed (Participants) | 10 | 10 | 10 | 10
Degrees/second | 35.2 (6.3) | 34.5 (9.3) | 37.2 (9.4) | 32.9 (10.8)

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Definition is same as ClinicalTrials.gov. Adverse events information were collected during data collection activities.
Groups:
- Upper Limb Absence Without Prosthesis: Individuals with upper limb loss not wearing their prosthesis.
- Upper Limb Absence With Prosthesis: Individuals with upper limb loss wearing their prosthesis.
Arm/Group | Healthy Controls With Arms Free | Upper Limb Absence Without Prosthesis | Healthy Controls With One Arm Bound | Upper Limb Absence With Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT04274218/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04274218/ICF_000.pdf